CLINICAL TRIAL: NCT05648513
Title: Evaluation of the Motivational Interview Teqhnique in Pregnant Women Who Are Hesitant in Applying Childhood Vaccines
Brief Title: The Motivational Interview Teqhnique in Pregnant Women Who Are Hesitant in Childhood Vaccines
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Balikesir University (Other)
Responsible Party: Principal Investigator, Selda Yoruk, Assoc.Dr., Balikesir University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: BAÜNSBF-ARSLAN-001
Record Dates: First submitted 2022-12-05; First posted 2022-12-13 (Actual); Last update posted 2022-12-13 (Actual); Status verified 2022-12

CONDITIONS: Vaccine Refusal; Pregnancy Related; Motivation
Keywords: Motivational interviewing, vaccine,vaccine hesitancy
MeSH Terms: conditions — Vaccination Refusal; Vaccination Hesitancy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Motivational Interview (Experimental): Parent Attitudes About Childhood Vaccines Survey (PACV) will be implemented to the pregnant women consulting to Atatürk City Hospital. Subjects with vaccine hesitancy will be randomly distributed to groups, and in this way, experimental (n=26) and control (n=26) groups will be formed. Routine antenatal monitoring will be kept with the control group. With the experimental group, on the other hand, motivational interviewing method will be implemented for 4 sessions of about 45 minutes each. Interviews will be held at 4 separate weekends, 1 session for each. Interviews will be performed via online means or face to face.
  Personal Details Form It is the survey form that includes such socio-demographic aspects of the participants as their ages and educational backgrounds, and their opinions about vaccines.
  Interventions: Behavioral: Motivational Interwiev
- Control Group (No Intervention): Control Group Experimental Group ( n=26 ) Routine antenatal monitoring will be kept with the control group. Routine antenatal monitoring Completion of motivational interviewing session Inspection of the vaccine card 1st and 2nd postnatal months and implementation of Parent Attitudes About Childhood Vaccines Survey (PACV) Personal Details Form It is the survey form that includes such socio-demographic aspects of the participants as their ages and educational backgrounds, and their opinions about vaccines.

INTERVENTIONS:
Behavioral: Motivational Interwiev — Parent Attitudes About Childhood Vaccines Survey (PACV) will be implemented to the patients consulting to Atatürk City Hospital. Subjects with vaccine hesitancy will be randomly distributed to groups, and in this way, experimental (n=26) and control (n=26) groups will be formed. Routine antenatal monitoring will be kept with the control group. With the experimental group, on the other hand, motivational interviewing method will be implemented for 4 sessions of about 45 minutes each. Interviews will be held at 4 separate weekends, 1 session for each. Interviews will be performed via online means or face to face.
  Arms: Motivational Interview

SUMMARY:
Vaccine hesitancy is defined by World Health Organization(WHO) "Vaccine Hesitancy Working Group" as a delay in acceptance or refusal of vaccines despite availability of vaccination services(MacDonald,2015). WHO listed "vaccine hesitancy" as one of the ten global health threats that require immediate solution in 2019(WHO, 2019). It was found out that the primary causes of vaccine hesitancy are the risk-benefit ratio concerns, including "concerns about the safety of vaccines" or "their potential side-effects", and secondary causes are the lack of information and awareness about vaccines and their importance and religious, cultural, social gender and socioeconomic perceptions of vaccination(Lark et al., 2018).It is estimated in social studies that the prevalence of vaccine hesitancy is about 25-70% in the top-ranking France, 15% in Switzerland and 19% in Canada(Ward et al.,2019; Shen and Dubey,2019). In the case of pregnant women, on the other hand, childhood vaccine hesitancy has been detected to vary between 6% and 12%(Mohd et al.,2017; Corben and Leask,2018).

There is a critical increase in the number of unvaccinated children in Turkey(Turkish Medical Association, 2018).Based on the data from Ministry of Health, number of families that refused to get their children vaccinated rose from 183 in 2011 to 12000 in 2016, and to 23600 in 2017(Turkish Medical Association, 2018).

Motivation is the probability of the individual to adopt, continue and adhere to the special strategies of change.MI is a directive and counselee-oriented approach, which is employed to help the patients explore and overcome the ambivalence/dilemma in adopting the behaviors that will enhance and improve their overall health.

Studies conducted in recent years have found out that motivational interviewing technique is actually effective in parents' acceptance of childhood vaccines. The main purpose of the MI technique is to explore the ambivalences of the target individuals and attain behavioral change by helping them overcome such ambivalences. This method is particularly useful with parents that are hesitant or ambivalent to get their children vaccinated, or those that fail to get them vaccinated. In MI, which focuses on the parents' concerns, questions and curiosities about the vaccines, the behavioral change takes place depending on the personal values of each individual. MI is a special means of aid to help individuals understand their problems and encourage them to take action(Danchin et al.,2017).

In order to enhance vaccination services, studies must be conducted on the issue of vaccine opposition and hesitancy of families, and underlying reasons must be revealed(Topçu et al.,2019; Akbaş,2020). Due to the fact that pregnancy and antenatal periods are the time spans when the first perspectives and beliefs about childhood vaccination are formed, these periods are particularly important for providing information pediatric vaccines. Determining the prevalence of vaccine opposition within the society, and monitoring it in upcoming years, as well as making programs on inspection and education, are assumed to be crucial in the struggle with vaccine hesitancy.

This study is particularly important as it will help eradicate vaccine hesitancy through using Motivational Interviewing (MI) method and revealing the ambivalent emotions about vaccine hesitancy in pregnant women.

DETAILED DESCRIPTION:
Main hypotheses/goal of the Study:

Hypothesis 0 Motivational Interviewing has no effect on vaccine hesitant pregnant women.

Hypothesis 1 Motivational Interviewing is effective on vaccine hesitant pregnant women.

Objective of the Study The study is a randomized experimental work conducted to analyze the effectiveness of Motivational Interviewing Method on pregnant women experiencing hesitancy about childhood vaccines.

Study Area:

The study will be conducted during March 2022-March 2023 in Balıkesir province. Balıkesir is located in the Southern Marmara sub-region, some of its land extending to Aegean Region. It is surrounded by Bursa and Kütahya to the east, Manisa and İzmir to the south, and Çanakkale to the west. The province is composed of 20 districs, 2 of them being the central districts. As per the 2020 findings of Turkish Statistical Institute (TUIK), it has a population of 1 240 285 people living in a total land area of 14 292 square kilometers. The main sources of income are agriculture and farming.

Planned data collection centers: Pregnant women visiting Atatürk Şehir Hastanesi (lit.Atatürk City Hospital) will be invited to participate in the research study.

Criteria to terminate the study:

The study will be terminated if it cannot be implemented due to reasons including disease and pandemic.

MATERIAL AND METHOD OF THE STUDY:

Population of the Study and sampling The population of the study comprises pregnant women residing in Balıkesir. Sampling size was calculated based on greater effect size in the intervention phase of the study. Using G-Power program, and given that α=0.05, power=0.95, effect size=0.80 according to bi-directional hypothesis, the sampling size was calculated to be 52 (control group: 26 and experimental group: 26)

Criteria for participation in the research study:

* Being pregnant for 28+ weeks,
* Experiencing hesitancy about childhood vaccines,
* Agreeing to participate in the study,
* Being literate,
* Having no communication disability,
* Volunteering to participate in the study,

Criteria for exclusion from the research study:

* Having high risk pregnancy
* Having psychiatric diseases
* Adolescent pregnancy
* Not accepting to participate in the study Data collection technique Parent Attitudes About Childhood Vaccines Survey (PACV) will be implemented to the patients consulting to Atatürk City Hospital. Subjects with vaccine hesitancy will be randomly distributed to groups, and in this way, experimental (n=26) and control (n=26) groups will be formed. Routine antenatal monitoring will be kept with the control group. With the experimental group, on the other hand, motivational interviewing method will be implemented for 4 sessions of about 45 minutes each. Interviews will be held at 4 separate weekends, 1 session for each. Interviews will be performed via online means or face to face.

Implementation Sessions of Motivational Interviewing Method is presented in Table 1 and Flowchart of the Study is Presented in Figure 1.

Table 1. Implementation Sessions of Motivational Interviewing Method

Sessions Contents

1. st Session (Week 1) - Acquaintance

   * Informing the individual about the interview (frequency/duration)
   * Revealing the rate of knowledge and attitudes of the individuals about vaccination
   * Identifying the reasons of vaccine hesitancy
   * Providing required information about vaccines
2. nd Session (Week 2) -Evaluation of the previous session

   * Reinforcement of motivation
   * Implementation of significance and reliability scale
   * Revealing the dilemma about vaccines
3. rd Session (Week 3) -Evaluation of the previous session

   * Reinforcement of motivation
   * Implementation of bidirectional decision balance
   * Evaluation of the "change" speech of the subject
   * If the change speech is evident, drafting transformation plan
4. th Session (Week 4) -Evaluation of the previous session

   * If ambivalence continues with the subject, speech on vaccination and stress on the importance of self- control
   * Reviewing the change plan, if it has been drawn up in previous session
   * Reinforcement of the sustainability of attained changes
   * Evaluation

Figure 1. Flow Chart of the Study

* Identification of pregnant women with vaccine hesitation (n=52)

Randomization (n=52)

* ↘ Control Group Experimental Group ( n=26 ) (n=26)

  * ↓ ↓ Routine antenatal monitoring Completion of motivational interviewing session
  * ↓ ↓ Inspection of the vaccine card 1st and 2nd postnatal months and implementation of Parent Attitudes About Childhood Vaccines Survey (PACV)

Personal Details Form It is the survey form that includes such socio-demographic aspects of the participants as their ages and educational backgrounds, and their opinions about vaccines.

Parent Attitudes About Childhood Vaccines Survey (PACV) It is a 10-point Likert scale; points 1-5 indicating hesitant response, points 6 and 7 uncertain response, and points 8-10 unhesitant response. Hesitant responses are assigned a 2, 'don't know or not sure' a 1, and non-hesitant responses a 0. After attributing points for each item, item scores are summed to obtain a total raw score. The total raw score was then converted to a scale ranging from 0 (least hesitant) to 100 (most hesitant), using simple linear transformation, Parents with a converted score ≥ 50 are identified as vaccine hesitant parents, while those with a converted score < 50 are identified as non-hesitant parents (Mutlu, 2021).

Variables of the Research Study Dependent variable: Vaccine hesitancy scores of the participants Independent Variable: Sociodemographic aspects of the participants (age, education, income etc.), pregnancy-derived aspects (week of pregnancy, planned or unplanned pregnancy etc.), implementation of MI Data Analysis Data will be analyzed on computer environment using SPSS 25 package software. Statistical significance will be accepted if p<0.05. In statistical analysis of the data, frequency and percentage values will be used for nominal data, whereas medians and standard deviation values will be used for numerical data. Normal distribution of the data will be assessed through Kolmogorov-Smirnov test. Univariate analysis and multivariate analysis methods and chi square test will be used in comparison of the nominal values across the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Being pregnant for 28+ weeks,
* Experiencing hesitancy about childhood vaccines,
* Agreeing to participate in the study,
* Being literate,
* Having no communication disability,
* Volunteering to participate in the study,

Exclusion Criteria:

* Having high risk pregnancy
* Having psychiatric diseases
* Adolescent pregnancy
* Not accepting to participate in the study

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 52 (Estimated)
Dates: Start 2022-12-28 (Estimated); Primary Completion 2023-04-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
Administered childhood vaccine | 6 months
  Inspection of the vaccine card 1st and 2nd postnatal months and
Vaccine Hesitant Score | 6 months
  implementation of Parent Attitudes About Childhood Vaccines Survey (PACV)

CONTACTS AND LOCATIONS:
Locations (1):
- Balikesir University, Balıkesir, Turkey (Türkiye)